CLINICAL TRIAL: NCT04795531
Title: A 26-week Double Blinded, Multiregional, Trial Comparing the Effect and Safety of Once Weekly Insulin Icodec and Once Daily Insulin Degludec 100 Units/mL, Both in Combination With Non-insulin Anti-diabetic Drugs, in Insulin naïve Subjects With Type 2 Diabetes.
Brief Title: A Research Study to Compare Two Types of Insulin, a New Insulin, Insulin Icodec and an Available Insulin, Insulin Degludec, in People With Type 2 Diabetes Who Have Not Used Insulin Before (ONWARDS 3)
Acronym: ONWARDS 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN1436-4479; U1111-1247-5218 (Other: World Health Organization (WHO)); 2020-000472-37 (EudraCT Number)
Record Dates: First submitted 2021-03-10; First posted 2021-03-12 (Actual); Results first posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin icodec; insulin degludec

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Once weekly insulin icodec + once daily placebo (Experimental): Participants will get once daily and once weekly injections
  Interventions: Drug: Insulin icodec; Drug: Placebo insulin degludec
- Once weekly placebo and once daily insulin degludec (Experimental): Participants will get once daily and once weekly injections
  Interventions: Drug: Placebo insulin icodec; Drug: Insulin degludec

INTERVENTIONS:
Drug: Insulin icodec — You will get a pen for weekly injection and one for daily injection. One will be icodec 700 units/mL and the other will be placebo.
  Subcutaneously (under the skin) injections
  Arms: Once weekly insulin icodec + once daily placebo
Drug: Placebo insulin icodec — You will get a pen for weekly injection and one for daily injection. One will be insulin degludec 100 units/mL and the other will be placebo.
  Subcutaneously (under the skin) injections
  Arms: Once weekly placebo and once daily insulin degludec
Drug: Insulin degludec — You will get a pen for weekly injection and one for daily injection. One will be degludec 100 units/mL and the other will be placebo.
  Subcutaneously (under the skin) injections
  Arms: Once weekly placebo and once daily insulin degludec
Drug: Placebo insulin degludec — You will get a pen for weekly injection and one for daily injection. One will be icodec 700 units/mL and the other will be placebo.
  Subcutaneously (under the skin) injections
  Arms: Once weekly insulin icodec + once daily placebo

SUMMARY:
This study compares insulin icodec (a new insulin taken once a week) to insulin degludec (an insulin taken once daily which is already available on the market) in people with type 2 diabetes.

The study will look at how well insulin icodec taken weekly controls blood sugar compared to insulin degludec taken daily.

Participants will get their study medicine in an injection pen. Participants will get a pen for weekly injection and one for daily injection. One will be icodec or degludec and the other will be dummy medicine. The treatment participants get is decided by chance. Participants and the study staff will not know which active medicine they get.

The insulin is injected with a needle in a skin fold in the thigh. The study could last for about 8 months. Participants will have 13 clinic visits and 17 phone calls with the study doctor. At 8 clinic visits participants will have blood samples taken. At 4 clinic visits participants cannot eat or drink (except for water) for 8 hours before the visit.

Women cannot take part if pregnant, breast-feeding or plan to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged above or equal to 18 years at the time of signing informed consent.
* Diagnosed with T2D (type 2 diabetes) greater than or equal to 180 days prior to the day of screening.
* HbA1c (glycated haemoglobin) from 7.0-11.0% (53.0-96.7 mmol/mol) both inclusive at screening confirmed by central laboratory analysis.
* Insulin naïve. However, short term insulin treatment for a maximum of 14 days prior to the day of screening is allowed, as is prior insulin treatment for gestational diabetes.
* Stable daily dose(s) greater than or equal to 90 days prior to the day of screening of any of the following anti-diabetic drug(s) or combination regimen(s):

  a.) Any metformin formulations greater than or equal to 1500 mg or maximum tolerated or effective dose. b.) Any metformin combination formulations greater than or equal to 1500 mg or maximum tolerated or effective dose. c.) Any of the following oral anti-diabetic drug classes including combinations (greater than or equal to half of the maximum approved dose according to local label or maximum tolerated or effective dose).:Sulfonylureas - Meglitinides (glinides) - DPP-4 inhibitors - SGLT2 inhibitors - Thiazolidinediones - Alpha-glucosidase inhibitors - Oral combination products (for the allowed individual Oral Anti-diabetic Drugs (OADs)) - Oral or injectable GLP-1-receptor agonists
* Body mass index (BMI) below or equal to 40.0 kg/m^2.

Exclusion Criteria:

* Any episodes (as declared by the subject or in the medical records) of diabetic ketoacidosis within 90 days prior to the day of screening.
* Myocardial infarction, stroke, hospitalisation for unstable angina pectoris or transient ischaemic attack within 180 days prior to the day of screening.
* Chronic heart failure classified as being in New York Heart Association (NYHA) Class IV at screening.
* Anticipated initiation or change in concomitant medications (for more than 14 consecutive days) known to affect weight or glucose metabolism (e.g. treatment with orlistat, thyroid hormones, or corticosteroids).
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within the past 90 days prior to screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 588 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (93):
- United States (26):
  - Lakeview Clinical Research, LLC, Guntersville, Alabama
  - American Clinical Trials, Buena Park, California
  - Headlands Research California, LLC, Escondido, California
  - Valley Research, Fresno, California
  - First Valley Medical Group, Lancaster, California
  - Est Cst Inst for Rsrch,Jksnvil, Jacksonville, Florida
  - Palm Harbor Medical Associates, Palm Harbor, Florida
  - Metabolic Research Institute Inc, West Palm Beach, Florida
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Cotton-Oneill Diabetes and End, Topeka, Kansas
  - Arcturus Healthcare, PLC, Troy, Michigan
  - Southgate Medical Group, LLP, West Seneca, New York
  - Physician's East Endocrinology, Greenville, North Carolina
  - Accellacare, Wilmington, North Carolina
  - Diab & Endo Assoc of Stark Co, Canton, Ohio
  - Providence Health Partners Ctr, Dayton, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Intend Research, Norman, Oklahoma
  - Hillcrest Clinical Research, Simpsonville, South Carolina
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - UT Southwestern Med Cntr, Dallas, Texas
  - PrimeCare Medical Group, Houston, Texas
  - Texas Diab & Endo, P.A., Round Rock, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - Chrysalis Clinical Research, St. George, Utah
  - Rainier Clin Res Ctr Inc, Renton, Washington
- Argentina (4):
  - STAT Research, Buenos Aires
  - Centro de Investigación Clínica, CABA
  - Medical Center of Diabetes and Nutrition, CABA
  - Instituto de Clínica Médica y Diabetes, Mendoza
- Austria (5):
  - Universitätsklinik für Innere Medizin Graz, Graz
  - Universitätsklinik für Innere Medizin, Graz
  - Barmh. Brüder Linz, Konventspital, Linz
  - Gesundheitszentrum Hetzendorf, Vienna
  - Hanusch-Krankenhaus, Wien, Vienna
- Brazil (4):
  - Quanta Diagnóstico Nuclear / Medicina Nuclear Alto da XV, Curitiba, Paraná
  - Centro de Diabetes Curitiba, Curitiba, Paraná
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul Ltda., Porto Alegre, Rio Grande do Sul
  - CPQuali Pesquisa Clínica Ltda, São Paulo, São Paulo
- Canada (15):
  - Commonwealth Medical Clinic, Mount Pearl, Newfoundland and Labrador
  - Eastern Health Authority, St. John's, Newfoundland and Labrador
  - LMC Diabetes & Endocrinology (Barrie), Barrie, Ontario
  - LMC ClinRsrh Inc.Brampton, Brampton, Ontario
  - LMC (Thornhill), Concord, Ontario
  - LMC Endo Ctr (Etobicoke) Ltd, Etobicoke, Ontario
  - Western Univ. Cnt for Studies in Fam Med, London, Ontario
  - LMC Research Inc. Ottawa, Nepean, Ontario
  - Bluewater Clin Res Group,Inc, Sarnia, Ontario
  - Centricity Research LMC, Toronto, Ontario
  - Dr. Anil K Gupta Medicine Professional Corporation, Toronto, Ontario
  - ViaCar Recherche Clinique Inc, Brossard, Quebec
  - Clinique de Recherche Medpharmgene Inc., Montreal, Quebec
  - LMC Clin Rsrch Inc. (Montreal), Saint-Laurent, Quebec
  - Diex Recherche Victoriaville, Victoriaville, Quebec
- China (13):
  - Chinese People's Liberation Army General Hospital, Beijing, Beijing Municipality
  - Beijing Pinggu Hospital, Beijing, Beijing Municipality
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - Cangzhou People's Hospital, Cangzhou, Hebei
  - Harrison International Peace Hospital, Hengshui, Hebei
  - Changzhou No.2 People's Hospital, Yanghu Branch, Changzhou, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University_Nanjing, Nanjing, Jiangsu
  - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Jiangsu University_Zhenjiang, Zhenjiang, Jiangsu
  - Jinan Central Hospital, Ji'nan, Shandong
  - Shanghai Tenth People's Hsopital, Tongji University, Shanghai, Shanghai Municipality
  - Shanghai Fifth People's Hospital, Shanghai, Shanghai Municipality
  - General Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
- Czechia (6):
  - Edumed Broumov, Broumov
  - Diahelp - diabetologie, Pardubice
  - DIALINE s.r.o., Plzeň 3
  - Diabet2 s.r.o., Prague
  - EUC Klinika Praha a.s., Prague
  - Fledip s.r.o., Prague
- Denmark (4):
  - Aarhus Universitetshospital Diabetes og Hormonsygdomme, Aarhus N
  - Sydvestjysk Sygehus Esbjerg, Esbjerg
  - Steno Diabetes Center Cph_Steno Diabetes Center Cph, Hellerup
  - Hvidovre Hospital Endokrinologisk forsk. afs. 159, Hvidovre
- France (8):
  - Les Hopitaux de Chartres-Hopital Louis Pasteur, Le Coudray
  - Centre Hospitalier de Narbonne, Narbonne
  - Ap-Hp-Hopital Bichat-Claude Bernard-1, Paris
  - Centre Hospitalier Universitaire de Bordeaux-Hopital Haut Leveque-2, Pessac
  - Hospices Civils de Lyon-Hopital Lyon Sud-1, Pierre-Bénite
  - Centre Hospitalier Universitaire de Nantes-Hopital Nord Laennec-3, Saint-Herblain
  - Centre Hospitalier Universitaire de Toulouse-Hopital Rangueil-2, Toulouse
  - Centre de Recherche Clinique Portes Du Sud, Vénissieux
- Mexico (2):
  - Arechavaleta Granell María del Rosario, Guadalajara, Jalisco
  - Investigación Médica Sonora S.C., Hermosillo, Sonora
- Advanced Clinical Research LLC, Bayamón, Puerto Rico
- Taiwan (5):
  - Changhua Christian Hospital, Changhua
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Chi Mei Medical Center, Tainan
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Philis-Tsimikas A, Bajaj HS, Begtrup K, Cailleteau R, Gowda A, Lingvay I, Mathieu C, Russell-Jones D, Rosenstock J. Rationale and design of the phase 3a development programme (ONWARDS 1-6 trials) investigating once-weekly insulin icodec in diabetes. Diabetes Obes Metab. 2023 Feb;25(2):331-341. doi: 10.1111/dom.14871. Epub 2022 Oct 14. PMID 36106652
- [Derived] Philis-Tsimikas A, Krogsdahl Bache J, Fu A, Kellerer M, Salvesen-Sykes K, Bain SC. Insights on Hospitalisations from the Phase 3a ONWARDS 1-6 Trials of Once-Weekly Insulin Icodec. Diabetes Ther. 2025 Aug;16(8):1615-1631. doi: 10.1007/s13300-025-01745-4. Epub 2025 Jun 4. PMID 40465144
- [Derived] Riddell MC, Heller S, Carstensen L, Rocha TMP, Kehlet Watt S, Woo VC. The effect of once-weekly insulin icodec vs once-daily basal insulin on physical activity-attributed hypoglycaemia in type 2 diabetes: a post hoc analysis of ONWARDS 1-5. Diabetologia. 2025 Jul;68(7):1416-1422. doi: 10.1007/s00125-025-06414-6. Epub 2025 Apr 5. PMID 40186685
- [Derived] Li Y, Kar S, Li C, Liu M, Luan Z, Yuan G, Zhong X, Mu Y. Once-Weekly Insulin Icodec Versus Once-Daily Insulin Degludec in Insulin-Naive Chinese Participants with Type 2 Diabetes: A Post Hoc Analysis of ONWARDS 3. Diabetes Ther. 2025 Apr;16(4):685-699. doi: 10.1007/s13300-025-01701-2. Epub 2025 Feb 28. PMID 40016570
- [Derived] Lingvay I, Asong M, Desouza C, Gourdy P, Kar S, Vianna A, Vilsboll T, Vinther S, Mu Y. Once-Weekly Insulin Icodec vs Once-Daily Insulin Degludec in Adults With Insulin-Naive Type 2 Diabetes: The ONWARDS 3 Randomized Clinical Trial. JAMA. 2023 Jul 18;330(3):228-237. doi: 10.1001/jama.2023.11313. PMID 37354562

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 89 sites in 11 countries as follows (number of sites that screened participants/ number of sites that randomised participants): Argentina (4/4), Austria (3/3), Brazil (4/4), Canada (14/13), China mainland (13/13), Czech Republic (6/6), Denmark (4/4), France (9/8), Mexico (2/2), Taiwan (5/5), United States (28/27).
Pre-assignment Details: After randomisation participants continued their pre-trial non-insulin anti-diabetic background medication throughout the entire trial except for sulfonylureas and glinides, which had to be reduced at randomisation by approximately 50% at the discretion of the investigator.
Groups:
- Insulin Icodec: Participants were to receive once weekly subcutaneous (s.c.) injection of insulin icodec using PDS290 prefilled pen-injector at a starting dose of 70 units (U) and once weekly placebo for 26 weeks. The dose was then adjusted once weekly to reach the glycaemic target of 4.4-7.2 millimoles per liter (mmol/L) based on 3 pre-breakfast self-measured plasma glucose (SMPG) values measured on 2 previous days and on the day of the titration. If at least one pre-breakfast SMPG value was: < 4.4 mmol/L: dose reduced by 20 U; If the mean was: 4.4-7.2 mmol/L- no adjustment; > 7.2 mmol/L- dose increased by 20 U.
- Insulin Degludec: Participants were to receive once daily s.c. injection of insulin degludec using PDS290 prefilled pen-injector at a starting dose of 10 U and once daily placebo for 26 weeks. The dose was then adjusted once weekly to reach the glycaemic target of 4.4-7.2 millimoles per liter mmol/L based on 3 pre-breakfast values measured on 2 previous days and on the day of the titration. If at least one pre-breakfast SMPG value was: < 4.4 mmol/L: dose reduced by 3 U; If the mean was: 4.4-7.2 mmol/L- no adjustment; > 7.2 mmol/L- dose increased by 3 U.
Period: Overall Study
Arm/Group | Insulin Icodec | Insulin Degludec
Started | 294 | 294
Full Analysis Set (FAS) | 294 | 294
Safety Analysis Set (SAS) | 293 | 294
Treated | 293 | 294
Completed | 288 | 286
Not Completed | 6 | 8
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 2
Not completed — Death | 2 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomised participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Icodec | Insulin Degludec | Total
Number analyzed (Participants) | 294 | 294 | 588
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.70 (10.19) | 58.56 (9.74) | 58.13 (9.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 110 | 219
  Male | 185 | 184 | 369
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 76 | 88 | 164
  Not Hispanic or Latino | 203 | 190 | 393
  Unknown or Not Reported | 15 | 16 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 80 | 85 | 165
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 6 | 15
  White | 179 | 175 | 354
  More than one race | 11 | 11 | 22
  Unknown or Not Reported | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycated Haemoglobin (HbA1c)
Description: Change in HbA1c from baseline (week 0) to week 26 is presented. The outcome data is evaluated based on the in-trial observation period. The in-trial period started at randomisation and ended at the date of: the last direct participant-site contact, withdrawal for participants who withdrew their informed consent, the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e., possibly an unscheduled phone visit) and death for participants who died before any of the above.
Time Frame: Baseline (Week 0), Week 26
Population: Full analysis set (FAS) included all randomised participants.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Insulin Icodec | Insulin Degludec
Number analyzed (Participants) | 294 | 294
Percentage of HbA1c | -1.57 (0.05) | -1.36 (0.05)
Statistical Analysis 1: Comparison: Insulin Icodec vs Insulin Degludec; The response and change from baseline in response after 26 weeks are analysed using an analysis of covariance (ANCOVA) model with treatment, region and sulfonylureas (SU)/glinides use as fixed factors, and baseline response as covariate; Test type: Non-Inferiority — Non-inferiority of insulin icodec was considered confirmed if the upper limit of the two-sided 95% confidence interval (CI) for mean treatment difference (insulin icodec minus insulin degludec) was strictly below 0.3%; p < 0.0001, ANCOVA; Treatment difference = -0.21, 95% CI 2-sided [-0.34 to -0.08]

2. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change in FPG from baseline (week 0) to week 26 is presented. The outcome data was evaluated based on the in-trial observation period. The in-trial period started at randomisation and ended at the date of: the last direct participant-site contact, withdrawal for participants who withdrew their informed consent, the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e., possibly an unscheduled phone visit) and death for participants who died before any of the above.
Time Frame: Baseline (Week 0), Week 26
Population: Full analysis set (FAS) included all randomised participants. Overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | Insulin Icodec | Insulin Degludec
Number analyzed (Participants) | 284 | 290
millimoles per liter (mmol/L) | -3.01 (0.11) | -2.99 (0.11)

3. Secondary Outcome: Number of Severe Hypoglycaemic Episodes (Level 3)
Description: Number of severe hypoglycaemic episodes (level 3) is presented. Severe hypoglycaemia (level 3) is defined as hypoglycaemia with severe cognitive impairment requiring external assistance for recovery. The outcome data was evaluated based on the on-tratment period. The on-treatment period started at the date of first dose of trial product as recorded on the electronic case report form (eCRF), and ended at the first date of any of the following: The end of trial visit (V30), the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin (corresponding to 5 weeks after the end of the dosing interval for both treatment arms) and the end-date for the in-trial observation period. The on-treatment period represented the time period in which a participant was considered exposed to trial product.
Time Frame: From baseline (week 0) to week 31
Population: Safety analysis set (SAS) included all participants randomly assigned to trial treatment and who took at least 1 dose of trial product.
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec | Insulin Degludec
Number analyzed (Participants) | 293 | 294
Episodes | 0 | 2

4. Secondary Outcome: Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (< 3.0 mmol/L (54 Milligrams Per Deciliter [mg/dL]), Confirmed by Blood Glucose [BG] Meter)
Description: Number of clinically significant hypoglycaemic episodes (level 2) (less than [<] 3.0 millimoles per liter (mmol/L) (54 mg/dL), confirmed by BG meter) is presented. Clinically significant hypoglycaemia (level 2) is defined as plasma glucose value of less than 3.0 mmol/L (54 mg/dL) confirmed by BG meter. The outcome data was evaluated based on the on-treatment period. The on-treatment period started at the date of first dose of trial product as recorded on the electronic case report form (eCRF), and ended at the first date of any of the following: The end of trial visit (V30), the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin (corresponding to 5 weeks after the end of the dosing interval for both treatment arms) and the end-date for the in-trial observation period. The on-treatment period represented the time period in which a participant was considered exposed to trial product.
Time Frame: From baseline (week 0) to week 31
Population: as for outcome 3
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec | Insulin Degludec
Number analyzed (Participants) | 293 | 294
Episodes | 53 | 23

5. Secondary Outcome: Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (<3.0 mmol/L (54 mg/dL), Confirmed by BG Meter) or Severe Hypoglycaemic Episodes (Level 3)
Description: Number of clinically significant hypoglycaemic episodes (level 2) (less than 3.0 mmol/L) (54 mg/dL), confirmed by blood glucose [BG] meter) or severe hypoglycaemic episodes (level 3) is presented. Severe hypoglycaemia (level 3) is defined as hypoglycaemia with severe cognitive impairment requiring external assistance for recovery. Clinically significant hypoglycaemia (level 2) is defined as plasma glucose value of < 3.0 mmol/L (54 mg/dL) confirmed by BG meter. The outcome data was evaluated based on the on-treatment period. The on-treatment period started at the date of first dose of trial product as recorded on the electronic case report form (eCRF), and ended at the first date of any of the following: The end of trial visit (V30), the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin (corresponding to 5 weeks after the end of the dosing interval for both treatment arms) and the end-date for the in-trial observation period.
Time Frame: From baseline (week 0) to week 31
Population: as for outcome 3
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec | Insulin Degludec
Number analyzed (Participants) | 293 | 294
Episodes | 53 | 25

6. Secondary Outcome: Number of Severe Hypoglycaemic Episodes (Level 3)
Description: Number of severe hypoglycaemic episodes (level 3) is presented. Severe hypoglycaemia (level 3) is defined as hypoglycaemia with severe cognitive impairment requiring external assistance for recovery.
Time Frame: From baseline (week 0) to week 26
Population: as for outcome 3
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec | Insulin Degludec
Number analyzed (Participants) | 293 | 294
Episodes | 0 | 0

7. Secondary Outcome: Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (<3.0 mmol/L (54 mg/dL), Confirmed by BG Meter)
Description: Number of clinically significant hypoglycaemic episodes (level 2) (< 3.0 mmol/L (54 mg/dL), confirmed by BG meter) is presented. Clinically significant hypoglycaemia (level 2) is defined as plasma glucose value of less than (<) 3.0 mmol/L (54 mg/dL) confirmed by BG meter.
Time Frame: From baseline (week 0) to week 26
Population: as for outcome 3
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec | Insulin Degludec
Number analyzed (Participants) | 293 | 294
Episodes | 50 | 17

8. Secondary Outcome: Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (<3.0 mmol/L (54 mg/dL), Confirmed by BG Meter) or Severe Hypoglycaemic Episodes (Level 3)
Description: Number of clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL), confirmed by BG meter) or severe hypoglycaemic episodes (level 3) is presented. Severe hypoglycaemia (level 3) is defined as hypoglycaemia with severe cognitive impairment requiring external assistance for recovery. Clinically significant hypoglycaemia (level 2) is defined as plasma glucose value of less than (<) 3.0 millimoles per liter (mmol/L) (54 milligrams per deciliter [mg/dL]) confirmed by blood glucose (BG) meter.
Time Frame: From baseline (week 0) to week 26
Population: as for outcome 3
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec | Insulin Degludec
Number analyzed (Participants) | 293 | 294
Episodes | 50 | 17

9. Secondary Outcome: Change in Body Weight
Description: Change in body weight from baseline (week 0) to week 26 is presented. The outcome data was evaluated based on the in-trial observation period. The in-trial period started at randomisation and ended at the date of: the last direct participant-site contact, withdrawal for participants who withdrew their informed consent, the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e., possibly an unscheduled phone visit) and death for participants who died before any of the above.
Time Frame: Baseline (Week 0), Week 26
Population: Full analysis set included all randomised participants.
Measure: Least Squares Mean (Standard Error); unit: Kilograms (kg)
Arm/Group | Insulin Icodec | Insulin Degludec
Number analyzed (Participants) | 294 | 294
Kilograms (kg) | 2.77 (0.22) | 2.32 (0.24)

10. Secondary Outcome: Mean Weekly Insulin Dose
Description: Estimated mean weekly insulin dose during the last 2 weeks of treatment (from week 24 to week 26) is presented. The outcome data was evaluated based on the on-treatment period. The on-treatment period started at the date of first dose of trial product as recorded on the electronic case report form (eCRF), and ended at the first date of any of the following: The end of trial visit (V30), the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin (corresponding to 5 weeks after the end of the dosing interval for both treatment arms) and the end-date for the in-trial observation period. The on-treatment period represented the time period in which a participant was considered exposed to trial product.
Time Frame: From week 24 to week 26
Population: Full analysis set included all randomised participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units (U) of insulin
Arm/Group | Insulin Icodec | Insulin Degludec
Number analyzed (Participants) | 294 | 294
Units (U) of insulin | 204.28 [189.44 to 220.29] | 186.52 [173.06 to 201.02]

ADVERSE EVENTS:
Time Frame: From baseline (Week 0) to Week 31
Description: All presented adverse events (AEs) are treatment emergent. A treatment-emergent AE (TEAE) was defined as an AE that initiated or worsened on or after the date of first dose of study drug up to the end of the trial period (week 31). Results are based on the safety analysis set (SAS) which included all participants randomly assigned to trial treatment and who took at least 1 dose of trial product.
Arm/Group | Insulin Icodec | Insulin Degludec
All-Cause Mortality (participants affected / at risk) | 2/293 | 1/294
Serious Adverse Events (participants affected / at risk) | 15/293 | 15/294
Other Adverse Events (participants affected / at risk) | 52/293 | 29/294
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Icodec (N=293) | Insulin Degludec (N=294)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Aortic arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Retinopathy hypertensive (Eye disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Icodec (N=293) | Insulin Degludec (N=294)
COVID-19 (Infections and infestations) | 24 (24) | 14 (14)
Diabetic retinopathy (Eye disorders) | 15 (16) | 6 (7)
Influenza (Infections and infestations) | 15 (18) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/31/NCT04795531/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/31/NCT04795531/SAP_001.pdf